CLINICAL TRIAL: NCT02492594
Title: Optimized Diagnostics for Improved Therapy Stratification in Invasive Fungal Infections
Acronym: FUNGITECT
Status: Completed | Type: Observational
Sponsor: St. Anna Kinderkrebsforschung (Other)
Responsible Party: Sponsor
Other Study IDs: VB MD-AN-007-3D
Record Dates: First submitted 2015-05-28; First posted 2015-07-08 (Estimated); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Systemic Mycosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Material that is not analyzed immediately will be stored until end of the study.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pediatric patients with febrile neutropenia: Peripheral blood sampling - samples from 200 pediatric patients with severe immunosuppression and neutropenic fever will be analyzed
  Interventions: Other: Peripheral blood sampling
- Adult patients with febrile neutropenia: Peripheral blood sampling - samples from 200 adult patients with severe immunosuppression and neutropenic fever will be analyzed
  Interventions: Other: Peripheral blood sampling

INTERVENTIONS:
Other: Peripheral blood sampling — Peripheral blood samples will be taken at 3-5 defined timepoints during febrile neutropenia:
  * at the start of neutropenic fever
  * after 24 hours
  * after 48 hours
  * before the start of antimycotic therapy, if pertinent
  * at the end of antimycotic therapy, if pertinent

SUMMARY:
Invasive fungal infections (IFI) in immunocompromised patients pose a major challenge for diagnostics designed to permit timely onset of appropriate treatment. The aim of the current clinical-diagnostic studies, one in in pediatric and one in adult patients at high risk of IFI, is to test newly developed diagnostic approaches to invasive fungal infections in relation to established procedures. The studies will be performed in a prospective, blinded fashion, and represent a work package within the FUNGITECT grant supported by the European Commission. The studies will focus on analyses of blood-samples from patients with febrile neutropenia during treatment of acute leukaemia and other tumour entities, and patients undergoing allogeneic stem cell transplantation treated with intensive chemotherapy.

DETAILED DESCRIPTION:
Samples from immunosuppressed patients with febrile neutropenia (NP - defined as fever ≥ 38.5ºC and <500 ANC) will be taken:

* at the start of neutropenic fever
* after 24 hours
* after 48 hours
* before the start of antimycotic therapy, if pertinent
* at the end of antimycotic therapy, if pertinent

The results ot analyses by a panfungal PCR screening assay developed at our institution (European patent No 1960536) and methods newly developed during the FUNGITECT project will be compared with conventional methods for fungal diagnostics such as HR (High Resolution)-CT, serological testing, histology and fungal culture. Additionally, genomic approaches will be employed to investigate host- and pathogen-related factors of susceptibility, pathogenicity and antimycotic resistance.

ELIGIBILITY:
INCLUSION CRITERIA

Adult study:

* Patients between 18-90 years of age with high risk of invasive fungal infections
* signed informed consent

Pediatric study:

* patients between 0-18 years of age with high risk of invasive fungal infections
* signed informed consent

EXCLUSION CRITERIA

Adult study:

* pregnancy
* no consent

Pediatric study:

- no consent

Ages: 6 Months to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. Adult Patients between 18-90 years of age with high risk of invasive fungal infections (patients suffering from acute leukaemia and other tumour entities treated with intensive chemotherapy with neutropenic fever
  2. Pediatric patients between 0-18 years of age with high risk of invasive fungal infections ((patients suffering from acute leukaemia, patients undergoing allogeneic stem cell transplantation treated with intensive chemotherapy with neutropenic fever.
Sampling Method: Non-Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with fungal DNAmia (as indicator of fungal infection) detected by new methodologies described in the proposal | until the end of antifungal treatment (up to 6 weeks after the onset of febrile neutropenia)
  Invasive fungal diseases will be evaluated by developing improved diagnosis: technical validation of individual assays (PCR-based, NGS, and protein-based), validation of biomarkers in clinical specimens (MoAbs, proteinaceous infection markers) and optimized for time and parallel processing of samples by establishing a robust protocol to generate reproducible results, implementation of automated or semi-automated techniques and by use of defined quality control systems.
Frequency of individual fungal pathogens during febrile neutropenia in high risk patients | until the end of antifungal treatment (up to 6 weeks after the onset of febrile neutropenia)
  The frequency of invasive fungal disease in the paediatric and adult patient cohorts as well as in each individual patient will be elucidated.
Frequency of fungal pathogens resistant to commonly used antifungal agents | until the end of antifungal treatment (up to 6 weeks after the onset of febrile neutropenia)
  Progress and changes in healthcare practices provide opportunities for new and drug-resistant fungal pathogens emerging in hospital settings.

SECONDARY OUTCOMES:
Number of lethal fungal infections | until the end of antifungal treatment (up to 6 weeks after the onset of febrile neutropenia)
  Evaluation of potentially life-threatening fungal infections according to EORTC criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lion, Prof MD PhD MSc, Study Chair — St. Anna Kinderkrebsforschung
Locations (7):
- Austria (5):
  - Medical University of Vienna, Department of Internal Medicine I, Vienna
  - Hospital Hietzing, Vienna
  - Hanusch Krankenhaus, Vienna
  - Wilhelminenspital, Vienna
  - St. Anna Children's Hospital, Vienna
- Princess Máxima Center for pediatric oncology, Utrecht, Netherlands
- First Saint-Petersburg Pavlov State Medical University, Saint Petersburg, Russia

REFERENCES:
- [Result] Landlinger C, Preuner S, Baskova L, van Grotel M, Hartwig NG, Dworzak M, Mann G, Attarbaschi A, Kager L, Peters C, Matthes-Martin S, Lawitschka A, van den Heuvel-Eibrink MM, Lion T. Diagnosis of invasive fungal infections by a real-time panfungal PCR assay in immunocompromised pediatric patients. Leukemia. 2010 Dec;24(12):2032-8. doi: 10.1038/leu.2010.209. Epub 2010 Sep 30. PMID 20882044
- [Derived] Lucini C, Obrova K, Krickl I, Nogueira F, Kocmanova I, Herndlhofer S, Gleixner KV, Sperr WR, Frank T, Andrade N, Peters C, Engstler G, Dworzak M, Attarbaschi A, van Grotel M, van den Heuvel-Eibrink MM, Moiseev IS, Rogacheva Y, Zubarovskaya L, Zubarovskaya N, Pichler H, Lawitschka A, Koller E, Keil F, Mayer J, Weinbergerova B, Valent P, Lion T. Prevalence of fungal DNAemia mediated by putatively non-pathogenic fungi in immunocompromised patients with febrile neutropenia: a prospective cohort study. J Hematol Oncol. 2024 Aug 7;17(1):63. doi: 10.1186/s13045-024-01583-0. PMID 39113112
- See also: Link to the web page of the Children's Cancer Research Institute (St. Anna Kinderkrebsforschung), the sponsor of the study. — http://www.kinderkrebsforschung.at/